CLINICAL TRIAL: NCT04947488
Title: Evaluation of the Effects of Treatment With Bioarginin C on Physical Exhaustion , Systemic Inflammatory State and Endothelial Function in Adult Subjects Belonging to the Post-Covid Day Hospital
Brief Title: Evaluation of the Effects of Treatment With Bioarginin C in Adult Subjects Belonging to the Post-Covid Day Hospital
Acronym: BC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Matteo Tosato, Doctor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Bioarginina C
Record Dates: First submitted 2021-06-30; First posted 2021-07-01 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Fatigue Syndrome, Chronic; Inflammation
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bioarginina C (Active Comparator): vials based on L-arginine and liposomal vitamin C
  Interventions: Dietary Supplement: Bioarginina C
- Placebo (Placebo Comparator): vials without L-arginine and liposomal vitamin C
  Interventions: Dietary Supplement: Bioarginina C

INTERVENTIONS:
Dietary Supplement: Bioarginina C — Dietary supplement vials

SUMMARY:
Long Covid could be much more frequent than it is thought to be. Few dwell on the great problem represented by the post covid syndrome. The virus often leaves important marks on our body, and those who recover face problems of various kinds: chronic fatigue, shortness of breath, dry cough, headache, cognitive difficulties.

On the duration and resolution of this syndrome, now recognized as a highly debilitating condition, there are still no great answers: for this reason it is always important to emphasize that contracting Covid, even in a not serious form, still means exposing oneself to long-term risks that are still not well codified by the scientific community. Guidelines and more tools are expected to best assist these patients.

ELIGIBILITY:
Inclusion Criteria:

subjects with proven positivity to the molecular test for Sars-cov2 with demonstration of microbiological healing patients discharged from FPG or other hospital structures; or only contact in PS; or home management age: range 20-60 years Fatigue operationalized as an affirmative answer to item "7" (CES-D)

Exclusion Criteria:

Pharmacological therapies with possible interactions with the mechanisms / processes under study (e.g. antihypertensive drugs, cortisone drugs, NSAIDs, immunosuppressants, nitrates)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-06-18 (Actual); Primary Completion 2022-09-18 (Estimated); Study Completion 2022-11-18 (Estimated)

PRIMARY OUTCOMES:
6 minute walking test to evaluate Fatigue | 30 days
  Effect of Bioarginina C on the prolonged fatigue

CONTACTS AND LOCATIONS:
Locations (1):
- Barbara Maglione, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No